CLINICAL TRIAL: NCT04461340
Title: Efficacy and Safety of Sirolimus for Treating COVID-19 Infection
Brief Title: Efficacy and Safety of Sirolimus in COVID-19 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sirolimus in COVID 19
Record Dates: First submitted 2020-07-04; First posted 2020-07-08 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID 19
Keywords: sirolimus; COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: single-blinded randomized clinical trial in which participants will be randomly assigned to one of the study groups using block randomization with a ratio of 1:1.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 20 patients will receive sirolimus ( oral dose of 6 mg on day 1 followed by 2 mg daily for 9 days) plus national standard of care therapy against COVID 19
  Interventions: Drug: Sirolimus
- Group B (No Intervention): 20 patients will receive only national standard of care therapy against COVID 19

INTERVENTIONS:
Drug: Sirolimus — oral dose of 6 mg on day1 followed by 2 mg daily for 9 days
  Other Names: Rapamune
  Arms: Group A

SUMMARY:
This research is planned to illustrate the efficacy and safety of sirolimus as an adjuvant agent to the standard treatment protocol against COVID-19 infection

DETAILED DESCRIPTION:
In early December 2019, several pneumonia cases of unknown origin were observed in Wuhan (China). A novel enveloped RNA β coronavirus was isolated and named severe acute respiratory syndrome coronavirus 2 (SARSCoV- 2). The new virus rapidly spread across China and worldwide. On March 11th 2020, the World Health Organization (WHO) declared coronavirus disease 2019 (COVID-19) a pandemic. As of 1July 2020, COVID-19 has been confirmed in 10,357,662 individuals globally with deaths reaching 508,055 with a morality of 5.37%. Egypt has 68,311 confirmed cases and 2935 deaths.

The virus mainly spreads through respiratory droplets from infected patients. The clinical spectrum of COVID-19 infection ranges from asymptomatic forms to severe pneumonia requiring hospitalization and isolation in critical care units with the need of mechanical ventilation due to acute respiratory distress syndrome (ARDS). Main symptoms include fever, fatigue and dry cough. Common laboratory findings include lymphopenia and elevated lactate dehydrogenase levels. Platelet count is usually normal or mildly decreased. C reactive protein (CRP) and erythrocyte sedimentation rate (ESR) are usually increased while procalcitonin levels are normal and elevation of procalcitonin usually indicates secondary bacterial infection. Ferritin, D-dimer, and creatine kinase elevation is associated with severe disease. Chest computed tomographic scans show a typical pattern of bilateral patchy shadows or ground glass opacity.

Severe COVID-19 conditions are usually due to an aggressive inflammatory response known as "cytokine storm" that is characterized by the release of a large amount of pro-inflammatory cytokines. Lung injury, multiorgan failure, and unfavorable prognosis of severe COVID-19 infection have been attributed mainly to the cytokine storm state.

Many proinflammatory cytokines elevate in COVID-19 patients including interleukin (IL)-1, IL-6, IL-8, IL-10, tumor necrosis factor (TNF)-α and interferon( IFN)-Ȣ stimulating immune cells to invade sites of infection causing endothelial dysfunction, vascular damage, alveolar damage and ARDS. Cytokine storm has been reported in several viral infections including influenza H5N1 virus, influenza H1N1 virus, and the two coronaviruses highly related to COVID-19; "SARS-CoV" and "MERSCoV".

Currently, there is no vaccine and/or specific therapeutic drugs targeting the SARS-CoV-2. Hence, it remains a major challenge to decide what potential therapeutic regimens to prevent and treat severe COVID-19 infections. Effective vaccines are essential to combat against the extremely contagious SARS-CoV-2. Until we have specific vaccines or therapeutic drugs targeting SARS-CoV-2, "repurposed" drugs have been used to treat COVID-19 patients. At present, treatment of SARS-CoV-2 infection are mainly repurposing the available therapeutic drugs and based on symptomatic conditions. Considering ARDS, followed by secondary infections, antibiotics, antiviral therapy, systemic corticosteroids, and anti-inflammatory drugs (including anti-arthritis drugs) are often used in the treatment regimens. Neuraminidase inhibitors, RNA synthesis inhibitors, convalescent plasma, and traditional herbal medicines have also been utilized in the treatment of COVID 19. Nevertheless, the efficacy of these treatment regimens remains to be verified by appropriately designed clinical trials. Sirolimus, also known as rapamycin, is an immunosuppressant that is used to prevent organ transplant rejection by inhibiting mammalian target of rapamycin (mTOR) kinase. mTOR plays a key role in viral replication. In an in vitro experiment, sirolimus has been shown to affect PI3K/AKT/mTOR pathway which inhibited MERS-CoV activity. Studies of patients hospitalized with influenza can further shed light on the antiviral effect of sirolimus. In a randomized clinical trial conducted on 38 patients with confirmed H1N1 pneumonia and on mechanical ventilator support, a group treated with corticosteroids and 2 mg/day of sirolimus for 14 days (N=19) showed significantly better clinical outcomes compared with the group treated with corticosteroids only, including shorter median duration of ventilator used. Delayed oseltamivir plus sirolimus treatment in pH1N1-infected mouse model further suggested a significant association between the sirolimus treatment and improved outcomes. At least one in silico study identified sirolimus as one of the 16 potential candidates for treating COVID-19 patients based on data from other human coronavirus infections using network-based drug repurposing model.

ELIGIBILITY:
Inclusion Criteria:

* Adults (˃18 years) COVID-19 positive patients (confirmed by PCR).
* Moderate infection ( pneumonia ± leucopenia or lymphopenia ).

Exclusion Criteria:

* Severe or life threatening COVID infection: Severe disease is defined as: dyspnea, respiratory frequency ≥ 30/min, blood oxygen saturation ≤ 93%, partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or lung infiltrates > 50% within 24 to 48 hours. Life threatening disease is defined as: respiratory failure, septic shock, and/or multiple organ dysfunction or failure .
* Pregnant or lactating females.
* Participation in any investigational clinical study, other than observational, within the past 30 days; or plans to participate in such a study at any time from the day of enrollment until 30 days post-treatment in the current study.
* Allergy or hypersensitivity to sirolimus.
* Taking immunosuppressive drugs.
* Glomerular filtration rate (GFR) < 30 ml/min by CKD-EPI equation.
* liver cirrhosis .
* Decompensated heart failure.
* known active tuberculosis (TB) or history of incompletely treated TB.
* Uncontrolled systemic bacterial or fungal infections.
* Drugs that may affect sirolimus level: antifungals, diltiazem, verapamil, nicardipine, phenytoin, phenobarbital, rifampicin, carbamazepine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical recovery | 14-28 days
  The duration from start of treatment to normalization of pyrexia, respiratory rate ,O2 saturation and relief of cough that is maintained for at least 72 hours.
Viral clearance | 14 days
  Two successive negative COVID-19 PCR analysis tests 48-72 hours apart

SECONDARY OUTCOMES:
radiological lung extension | 14 days
  Evaluate the lung extension of pneumonia at day 14
drug adverse events | 28 days
  incidence and type of adverse events
28 day mortality | 28 day
  number of deaths to total number of patients
intensive care unit (ICU) admission rate | 28 days
  deteriorated patients who need admission to intensive care unit
Duration of hospital stay | 28 days
  duration from hospitalization to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; Ayman I Baess, MD, Study Chair — Associate professor; Heba M El weshahi, MD, Study Chair — professor; Nermine H Zakaria, MD, Study Chair — professor
Locations (1):
- Faculty of Medicine, Alexandria university, Egypt, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chan JF, Yuan S, Kok KH, To KK, Chu H, Yang J, Xing F, Liu J, Yip CC, Poon RW, Tsoi HW, Lo SK, Chan KH, Poon VK, Chan WM, Ip JD, Cai JP, Cheng VC, Chen H, Hui CK, Yuen KY. A familial cluster of pneumonia associated with the 2019 novel coronavirus indicating person-to-person transmission: a study of a family cluster. Lancet. 2020 Feb 15;395(10223):514-523. doi: 10.1016/S0140-6736(20)30154-9. Epub 2020 Jan 24. PMID 31986261
- [Background] Singhal T. A Review of Coronavirus Disease-2019 (COVID-19). Indian J Pediatr. 2020 Apr;87(4):281-286. doi: 10.1007/s12098-020-03263-6. Epub 2020 Mar 13. PMID 32166607
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Sun D, Li H, Lu XX, Xiao H, Ren J, Zhang FR, Liu ZS. Clinical features of severe pediatric patients with coronavirus disease 2019 in Wuhan: a single center's observational study. World J Pediatr. 2020 Jun;16(3):251-259. doi: 10.1007/s12519-020-00354-4. Epub 2020 Mar 19. PMID 32193831
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Lu H. Drug treatment options for the 2019-new coronavirus (2019-nCoV). Biosci Trends. 2020 Mar 16;14(1):69-71. doi: 10.5582/bst.2020.01020. Epub 2020 Jan 28. PMID 31996494
- [Background] Seto B. Rapamycin and mTOR: a serendipitous discovery and implications for breast cancer. Clin Transl Med. 2012 Nov 15;1(1):29. doi: 10.1186/2001-1326-1-29. PMID 23369283
- [Background] Kindrachuk J, Ork B, Hart BJ, Mazur S, Holbrook MR, Frieman MB, Traynor D, Johnson RF, Dyall J, Kuhn JH, Olinger GG, Hensley LE, Jahrling PB. Antiviral potential of ERK/MAPK and PI3K/AKT/mTOR signaling modulation for Middle East respiratory syndrome coronavirus infection as identified by temporal kinome analysis. Antimicrob Agents Chemother. 2015 Feb;59(2):1088-99. doi: 10.1128/AAC.03659-14. Epub 2014 Dec 8. PMID 25487801
- [Background] Wang CH, Chung FT, Lin SM, Huang SY, Chou CL, Lee KY, Lin TY, Kuo HP. Adjuvant treatment with a mammalian target of rapamycin inhibitor, sirolimus, and steroids improves outcomes in patients with severe H1N1 pneumonia and acute respiratory failure. Crit Care Med. 2014 Feb;42(2):313-21. doi: 10.1097/CCM.0b013e3182a2727d. PMID 24105455
- [Background] Jia X, Liu B, Bao L, Lv Q, Li F, Li H, An Y, Zhang X, Cao B, Wang C. Delayed oseltamivir plus sirolimus treatment attenuates H1N1 virus-induced severe lung injury correlated with repressed NLRP3 inflammasome activation and inflammatory cell infiltration. PLoS Pathog. 2018 Nov 13;14(11):e1007428. doi: 10.1371/journal.ppat.1007428. eCollection 2018 Nov. PMID 30422993
- [Background] Zhou Y, Hou Y, Shen J, Huang Y, Martin W, Cheng F. Network-based drug repurposing for novel coronavirus 2019-nCoV/SARS-CoV-2. Cell Discov. 2020 Mar 16;6:14. doi: 10.1038/s41421-020-0153-3. eCollection 2020. PMID 32194980